CLINICAL TRIAL: NCT07171762
Title: A Randomized Controlled Trial Comparing Intracanal Ozone Therapy and Conventional Irrigation on Oxidative Stress in Asymptomatic Apical Periodontitis
Brief Title: Effect of Ozone Use in Intracanal Irrigation on Oxidative Stress Level in Teeth With Asymptomatic Apical Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KEZBAN MELTEM ÇOLAK (Other)
Responsible Party: Sponsor-Investigator, KEZBAN MELTEM ÇOLAK, Professor of Endodontics,, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B.30.2.ATA.0.01.00/557
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Apical Periodontitis; Oxidative Stress
Keywords: Ozone Therapy; Endodontics; Oxidative Stress; Apical Periodontitis; Intracanal Irrigation; Antioxidant Status; Oxidant Status; Malondialdehyde (MDA); 8-Hydroxydeoxyguanosine (8-OHdG)
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups. The experimental group received ozone irrigation and the control group received saline irrigation during endodontic treatment. Oxidative stress markers were analyzed at multiple time points.
Who Masked: Participant
Masking Description: This study uses a single-blind design in which the participants are unaware of the intervention type (ozone or saline irrigation) they receive. The operator performing the root canal therapy is aware of the group assignment due to the nature of the intervention procedure. Outcome assessments are performed by the same clinician and are thus not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone Irrigation Group (Experimental): Participants in this arm will undergo root canal irrigation using ozonated water instead of conventional irrigants. Ozonated water is generated using a medical ozone generator (Ozonytron XP) and applied passively into the canal space. The aim is to evaluate its effect on oxidative stress markers such as TAS, TOS, MDA, and 8-OHdG in periapical fluid collected before and after irrigation. The irrigation protocol includes passive delivery with 30G side-vented needles following initial canal shaping. No sodium hypochlorite or EDTA is used in this group. This arm is designed to assess the biological impact of ozonated water as an alternative disinfection protocol in asymptomatic apical periodontitis.
  Interventions: Device: Ozonytron XP
- Saline Irrigation Group (Control) (Active Comparator): Participants in this group will receive conventional root canal irrigation using sterile saline (0.9% NaCl) solution. This irrigation is delivered passively into the canal space after instrumentation, using 30G side-vented irrigation needles. No active chemical disinfectant such as NaOCl or EDTA is used in this arm. Periapical fluid samples will be collected before and after irrigation, and analyzed for oxidative stress markers (TAS, TOS, MDA, and 8-OHdG). This group serves as a control to compare the biological effects of ozonated water irrigation in asymptomatic apical periodontitis cases
  Interventions: Other: Physiological saline solution (0.9% NaCl)

INTERVENTIONS:
Device: Ozonytron XP — This intervention involves the use of ozonated water as a final irrigation solution during root canal treatment in teeth diagnosed with asymptomatic apical periodontitis. Following standard chemomechanical preparation, ozonated water is delivered into the root canal system using a 30-gauge side-vented needle. The aim is to assess the biochemical changes in periapical tissues by evaluating oxidative stress markers (TAS, TOS, MDA, 8-OHdG) in the apical fluid samples collected before and after irrigation. The ozonated water is generated via a medical-grade ozone generator, and its application is designed to minimize cytotoxicity while maximizing antimicrobial and oxidative stress modulation properties. The outcomes are compared to a control group receiving saline irrigation under identical procedural conditions.
  Arms: Ozone Irrigation Group
Other: Physiological saline solution (0.9% NaCl) — Physiological saline solution (0.9% NaCl) was used as the final irrigation agent in root canal treatment.Saline Irrigation Group (Control)
  Arms: Saline Irrigation Group (Control)

SUMMARY:
This clinical study aims to investigate the oxidative stress-related effects of ozone irrigation in patients with asymptomatic apical periodontitis undergoing root canal treatment. A total of 60 patients who meet the inclusion criteria will be randomly assigned into two groups using an online randomization tool: an ozone irrigation group and a saline irrigation (control) group. The primary objective is to assess the biochemical effects of ozone therapy on oxidative stress markers in periapical interstitial fluid, including but not limited to TAS, TOS, MDA, and 8-OHdG, by using ELISA kits.

After routine canal preparation and initial irrigation protocol (NaOCl-EDTA-NaOCl), baseline periapical fluid samples will be collected using standardized sterile paper points. Following this, experimental irrigation will be applied: ozone water in the study group and saline solution in the control group. Second periapical fluid samples will be collected immediately after this procedure. Subsequently, calcium hydroxide dressing will be placed into the canals, and the patients will be recalled after one week. At the second visit, after removal of the intracanal medicament, a third sample will be collected from each patient.

Ethical approval was obtained from the Non-Interventional Clinical Research Ethics Committee of Atatürk University Faculty of Medicine. The results of this study are expected to contribute to the understanding of ozone therapy as a biocompatible and effective disinfection agent in endodontic procedures and to provide insights into its role in modulating oxidative stress within the periapical environment.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the effect of ozone irrigation on oxidative stress levels in teeth diagnosed with asymptomatic apical periodontitis. Apical periodontitis, characterized by inflammation of periapical tissues in response to persistent root canal infection, often progresses silently and can affect long-term endodontic success. In recent years, ozone therapy has gained attention due to its strong antimicrobial, anti-inflammatory, and tissue-regenerative properties. This study evaluates whether ozone irrigation during endodontic treatment can modulate oxidative stress biomarkers more effectively than traditional saline irrigation.

Study Objective

The primary aim is to compare oxidative stress marker levels (TAS, TOS, MDA, and 8-OHdG) in periapical fluid samples following ozone versus saline irrigation

. Study Design and Participants

A total of 60 patients aged between 18-65, each diagnosed with a single-rooted tooth exhibiting asymptomatic apical periodontitis, were included based on strict inclusion/exclusion criteria. Patients with systemic disease, recent antibiotic use, or periodontal involvement were excluded. Randomization was conducted via [www.randomizer.org](http://www.randomizer.org) to allocate participants into two groups (n=30 each):

Group A: Ozone irrigation group Group B: Saline (control) irrigation group

Each patient provided written informed consent, and the study received ethical approval from the Atatürk University Non-Interventional Clinical Research Ethics Committee (Decision No: B.30.2.ATA.0.01.00/557, Date: 27.09.2024).

Endodontic Procedure and Sampling Phases

After local anesthesia (2% articaine with 1:100,000 epinephrine) and rubber dam isolation, standardized root canal preparation was performed using rotary NiTi systems. During shaping, 2.5% NaOCl was used for initial irrigation. Final irrigation protocol common to both groups involved:

* 5 mL of 2.5% NaOCl
* 5 mL of 17% EDTA
* 5 mL of 2.5% NaOCl again

All irrigations were performed using 30-gauge side-vented needles.

Periapical Fluid Sampling Points

Sampling was done using sterile paper points inserted 2 mm beyond the apex, each held for 1 minute, and repeated with 3 paper points per canal. Each sample was stored in PBS-filled, coded Eppendorf tubes at -80°C.

Sample 1 (Baseline):

Collected immediately after final irrigation.

Sample 2 (After group-specific irrigation):

Group A received 5 mL of ozone water irrigation. Group B received 5 mL of sterile saline irrigation.

Samples were collected again using the same protocol.

Sample 3 (Post-medication):

Calcium hydroxide was placed as intracanal medicament. Patients were recalled after 7 days, Ca(OH)₂ was removed, and a third sample was obtained.

Laboratory Analysis

All samples were stored at -80°C until biochemical analysis. The oxidative stress markers were quantified using commercial ELISA kits according to manufacturer protocols.

Outcome Measures

Change in oxidative stress levels (TAS, TOS, MDA, 8-OHdG) at three time points.

Significance of the Study

This is the first known randomized clinical trial to assess the influence of ozone irrigation on oxidative stress biomarkers in periapical fluid. Given the potential of oxidative stress to affect tissue healing and inflammation, understanding the biochemical impact of ozone could offer novel insight into improving endodontic outcomes, especially in cases where apical healing is critical.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must be between 18 and 65 years of age 2. Single-rooted, asymptomatic apical periodontitis with necrotic teeth 3. Teeth with periapical lesion size classified as score 3 or 4 according to the Orstavik classification 4. Periapical Assessment Index (PAI) of 2 or higher 5. Patients with ASA I status

Exclusion Criteria

1. Teeth with multiple roots
2. Patients with ASA II or higher
3. Pregnant women or those suspected of being pregnant
4. Patients with a history of allergies
5. Teeth with excessive material loss where a rubber dam cannot be applied
6. Teeth with root fractures or an open apex
7. Teeth that have previously undergone root canal treatment
8. Presence of canal curvature greater than Schilder 25°,
9. Patients with generalized periodontitis,
10. Presence of a periodontal pocket greater than 3mm in the relevant tooth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in oxidative stress biomarkers in periapical fluid following ozone or saline irrigation | From baseline to 7 days after treatment
  The primary outcome is the quantitative change in oxidative stress markers including Total Antioxidant Status (TAS), Total Oxidant Status (TOS), Malondialdehyde (MDA), and 8-Hydroxy-2'-deoxyguanosine (8-OHdG) in periapical fluid. Measurements are taken at three time points:
  Immediately after canal preparation and final irrigation (ozonated water or saline), After application of the irrigant (ozonated water in the test group, saline in the control group), One week later, following the removal of calcium hydroxide medication. Samples are collected using sterile paper points and analyzed using ELISA and Western blot techniques. The purpose is to evaluate the antioxidant and oxidative stress responses to ozonated water compared to saline.

CONTACTS AND LOCATIONS:
Overall Officials: Kezban Meltem Çolak, Prof.Dr., Principal Investigator — ATATURK UNIVERSITY, FACULTY of DENTISTRY, Department of ENDODONTICS
Locations (1):
- ATATURK UNIVERSITY, FACULTY of DENTISTRY, Department of ENDODONTICS, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azarpazhooh A, Limeback H. The application of ozone in dentistry: a systematic review of literature. J Dent. 2008 Feb;36(2):104-16. doi: 10.1016/j.jdent.2007.11.008. Epub 2007 Dec 31. PMID 18166260
- [Background] Kazancioglu HO, Kurklu E, Ezirganli S. Effects of ozone therapy on pain, swelling, and trismus following third molar surgery. Int J Oral Maxillofac Surg. 2014 May;43(5):644-8. doi: 10.1016/j.ijom.2013.11.006. Epub 2013 Dec 11. PMID 24332588
- [Background] Nagayoshi M, Fukuizumi T, Kitamura C, Yano J, Terashita M, Nishihara T. Efficacy of ozone on survival and permeability of oral microorganisms. Oral Microbiol Immunol. 2004 Aug;19(4):240-6. doi: 10.1111/j.1399-302X.2004.00146.x. PMID 15209994
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18166260/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15209994/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24332588/
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/18166260/